CLINICAL TRIAL: NCT02386839
Title: Long-term Outcome of Children Enrolled in Study ROPP-2008-01 Previously Treated With rhIGF-1/rhIGFBP-3 for the Prevention of Retinopathy of Prematurity (ROP) or Who Received Standard Neonatal Care
Brief Title: Long-term Safety and Efficacy Outcome Study Comparing Children Previously Enrolled in Study ROPP-2008-01 for the Prevention of Retinopathy of Prematurity (ROP)
Acronym: PEDAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP607-201; 2014-003556-31 (EudraCT Number)
Record Dates: First submitted 2015-03-04; First posted 2015-03-12 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Insulin-Like Growth Factor I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Antecedent Standard of Care (Experimental): Participants who were treated with standard neonatal care in study ROPP-2008-01 (NCT01096784) were enrolled in this group for assessment of rhIGF-1/rhIGFBP-3 long-term efficacy and safety outcomes.
  Interventions: Drug: rhIGF-1/rhIGFBP-3
- Antecedent rhIGF-1/rhIGFBP-3 (Experimental): Participants who were treated with rhIGF-1/rhIGFBP-3 in study ROPP-2008-01 (NCT01096784) were enrolled in this group for assessment of rhIGF-1/rhIGFBP-3 long-term efficacy and safety outcomes.
  Interventions: Drug: rhIGF-1/rhIGFBP-3

INTERVENTIONS:
Drug: rhIGF-1/rhIGFBP-3 — Participants who received "rhIGF-1/rhIGFBP-3" in study ROPP-2008-01 (NCT01096784) will be enrolled to this study. No investigational product will be administered in this study.
  Other Names: Mecasermin rinfabate

SUMMARY:
The main purpose of this study is to evaluate the long-term efficacy and safety outcomes following short-term exposure to rhIGF-1/rhIGFBP-3 versus standard neonatal care in Study ROPP-2008-01 (NCT01096784).

DETAILED DESCRIPTION:
Long-term Safety and Efficacy Outcome Study Comparing Children Previously Enrolled in Study ROPP-2008-01 for the Prevention of Retinopathy of Prematurity (ROP)

ELIGIBILITY:
Inclusion Criteria:

* Participant was randomized in Study ROPP-2008-01 Section D (NCT01096784).
* Participants parent or legally authorized representative(s) must provide written informed consent prior to performing any study-related activities. Study-related activities are any procedures that would not have been performed during normal management of the participant.

Exclusion Criteria:

* Any other condition or therapy that, in the Investigator's opinion, may pose a risk to the Participant or interfere with the participants ability to be compliant with this protocol or interfere with the interpretation of results.
* The participant or participants parent or legally authorized representative(s) is unable to comply with the protocol as determined by the Investigator.

Ages: 40 Weeks to 108 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (16):
- United States (4):
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - Vidant Medical Center, Greenville, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Wisconsin - Madison, Madison, Wisconsin
- Italy (4):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Giannina Gaslini-Istituto Pediatrico di Ricovero e, Genova
  - University of Padua, Padua
  - Policlinico Universitario Agostino Gemelli, Roma
- VU Medical Center, Amsterdam, Netherlands
- Ginekologiczno-Położniczy Szpital Kliniczny Uniwersytetu Medycznego w Poznan, Poznan, Poland
- Sweden (2):
  - Skanes Universitetssjukhus Lund, Lund
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- United Kingdom (4):
  - Addenbrookes Hospital, Cambridge
  - St Peter's Hospital, Chertsey
  - Alder Hey Childrens Hospital, Liverpool
  - UCL EGA Institute for Women's Health, London

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 sites from 26 March 2015 (first participant first visit) to 28 September 2021 (last participant last visit).
Pre-assignment Details: A total of 76 participants who previously treated with rhIGF 1/rhIGFBP-3 or Standard Neonatal Care in ROPP-2008-01 (NCT01096784) study were enrolled in this long-term safety and efficacy study.
Groups:
- Antecedent Standard of Care: Participants who were treated with standard neonatal care in study ROPP-2008-01 (NCT01096784).
- Antecedent rhIGF-1/rhIGFBP-3: Participants who were treated with rhIGF-1/rhIGFBP-3 in study ROPP-2008-01 (NCT01096784).
Period: Overall Study
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Started | 36 | 40
Completed | 20 | 25
Not Completed | 16 | 15
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Lost to Follow-up | 4 | 4
Not completed — Other (Site Terminated by Sponsor) | 1 | 0
Not completed — Other (Covid 19 Pandemic) | 0 | 1
Not completed — Other (unspecified) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled set included all participants for whom written informed consent was obtained for this long-term outcome study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3 | Total
Number analyzed (Participants) | 36 | 40 | 76
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — The age reported here is the corrected age. Corrected Age (weeks) was defined as Chronological Age (weeks) - 40 + Gestational Age (weeks) in this study.
  Weeks | 7.15 (5.622) | 6.73 (6.224) | 6.93 (5.911)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 23 | 26 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 13 | 19
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 26 | 34 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Visual Acuity as Assessed by an Age-appropriate Method at 6 Months Corrected Age (CA)
Description: Standard age-appropriate methods were used to assess visual acuity (how well a participant sees at different distances) with teller acuity cards, LEA symbols test and Charts. It was categorized as following: normal (measurable acuity >= 20/40 or >= 15 cycles/degree); below normal (20/200 <= measurable acuity < 20/40 or 3 cycles/degree <= measurable acuity < 15 cycles/degree); poor (measurable acuity <= 20/200 or <= 3 cycles/degree). Corrected Age (weeks) was defined as Chronological Age (weeks) - 40 + Gestational Age (weeks) in this study.
Time Frame: At 6 Months CA
Population: Enrolled set included all participants for whom written informed consent was obtained for this long-term outcome study. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 27 | 34
Participants
  Participants With Right Eye: number analyzed (Participants) | 24 | 32
  Participants With Right Eye: Normal | 0 | 0
  Participants With Right Eye: Below Normal | 12 | 19
  Participants With Right Eye: Poor | 12 | 13
  Participants With Left Eye: number analyzed (Participants) | 21 | 32
  Participants With Left Eye: Normal | 0 | 0
  Participants With Left Eye: Below Normal | 14 | 18
  Participants With Left Eye: Poor | 7 | 14
  Participants With Both Eyes: Normal | 0 | 0
  Participants With Both Eyes: Below Normal | 18 | 25
  Participants With Both Eyes: Poor | 9 | 9

2. Primary Outcome: Number of Participants With Visual Acuity as Assessed by an Age-appropriate Method at 12 Months CA
Description: as for outcome 1
Time Frame: At 12 Months CA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 24 | 36
Participants
  Participants With Right Eye: number analyzed (Participants) | 21 | 32
  Participants With Right Eye: Normal | 0 | 1
  Participants With Right Eye: Below Normal | 21 | 26
  Participants With Right Eye: Poor | 0 | 5
  Participants With Left Eye: number analyzed (Participants) | 21 | 32
  Participants With Left Eye: Normal | 0 | 1
  Participants With Left Eye: Below Normal | 20 | 25
  Participants With Left Eye: Poor | 1 | 6
  Participants With Both Eyes: Normal | 0 | 1
  Participants With Both Eyes: Below Normal | 23 | 33
  Participants With Both Eyes: Poor | 1 | 2

3. Primary Outcome: Number of Participants With Visual Acuity as Assessed by an Age-appropriate Method at 20 Months CA
Description: as for outcome 1
Time Frame: At 20 Months CA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 33
Participants
  Participants With Right Eye: number analyzed (Participants) | 19 | 29
  Participants With Right Eye: Normal | 0 | 2
  Participants With Right Eye: Below Normal | 17 | 23
  Participants With Right Eye: Poor | 2 | 4
  Participants With Left Eye: number analyzed (Participants) | 20 | 29
  Participants With Left Eye: Normal | 0 | 1
  Participants With Left Eye: Below Normal | 18 | 24
  Participants With Left Eye: Poor | 2 | 4
  Participants With Both Eyes: Normal | 0 | 1
  Participants With Both Eyes: Below Normal | 20 | 30
  Participants With Both Eyes: Poor | 3 | 2

4. Primary Outcome: Number of Participants With Visual Acuity as Assessed by an Age-appropriate Method at 24 Months CA
Description: as for outcome 1
Time Frame: At 24 Months CA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 33
Participants
  Participants With Right Eye: number analyzed (Participants) | 20 | 31
  Participants With Right Eye: Normal | 0 | 2
  Participants With Right Eye: Below Normal | 17 | 25
  Participants With Right Eye: Poor | 3 | 4
  Participants With Left Eye: number analyzed (Participants) | 20 | 28
  Participants With Left Eye: Normal | 0 | 2
  Participants With Left Eye: Below Normal | 17 | 24
  Participants With Left Eye: Poor | 3 | 2
  Participants With Both Eyes: Normal | 1 | 5
  Participants With Both Eyes: Below Normal | 19 | 24
  Participants With Both Eyes: Poor | 3 | 4

5. Primary Outcome: Number of Participants With Visual Acuity as Assessed by an Age-appropriate Method at 4.75 Years CA
Description: as for outcome 1
Time Frame: At 4.75 Years CA
Population: Enrolled set included all participants for whom written informed consent was obtained for this long-term outcome study. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 15 | 18
Participants
  Participants With Right Eye: Normal | 11 | 15
  Participants With Right Eye: Below Normal | 4 | 3
  Participants With Right Eye: Poor | 0 | 0
  Participants With Left Eye: Normal | 11 | 14
  Participants With Left Eye: Below Normal | 4 | 4
  Participants With Left Eye: Poor | 0 | 0
  Participants With Both Eyes: Normal | 10 | 17
  Participants With Both Eyes: Below Normal | 5 | 1
  Participants With Both Eyes: Poor | 0 | 0

6. Primary Outcome: Number of Participants With Visual Acuity as Assessed by an Age-appropriate Method at 5 Years CA
Description: as for outcome 1
Time Frame: At 5 Years CA
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 14 | 17
Participants
  Participants With Right Eye: Normal | 9 | 11
  Participants With Right Eye: Below Normal | 5 | 6
  Participants With Right Eye: Poor | 0 | 0
  Participants With Left Eye: Normal | 8 | 11
  Participants With Left Eye: Below Normal | 6 | 6
  Participants With Left Eye: Poor | 0 | 0
  Participants With Both Eyes: Normal | 9 | 11
  Participants With Both Eyes: Below Normal | 5 | 6
  Participants With Both Eyes: Poor | 0 | 0

7. Primary Outcome: Number of Participants With Oculomotor Examination (Motility) and Ocular Alignment (Assessed by Corneal Light Reflex and Cover Test) at 12 Months CA
Description: Ocular alignment was assessed in primary gaze by comparing the position of the corneal light reflection in left eye and right eye (corneal light reflection assessment). Presence or absence of strabismus was recorded in primary gaze and in as many of the 9 positions of gaze as feasible with the cover test assessment of refixation movement. Extraocular muscle over action or deficiency was recorded. Ocular motility referred to eye movements governed by the 6 extraocular muscles in each eye. It was assessed by examiner observation of the participants ability to abduct, adduct, supra, and inferoduct each eye. Ocular alignment and motility included the presence or absence of strabismus (classified as Esotropia [inward turn of the eye], Exotropia [outward turn of the eye], Hypertropia [upward turn of the eye], Hypotropia [downward turn of the eye]) was recorded. Number of participants with combined data for ocular alignment and oculomotor examination (motility) at 12 months CA were reported.
Time Frame: At 12 Months CA
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 25 | 36
Participants
  Participants with Esotropia: Presence | 1 | 4
  Participants with Esotropia: Absence | 24 | 32
  Participants with Exotropia: Presence | 0 | 0
  Participants with Exotropia: Absence | 25 | 36
  Participants with Hypertropia: Presence | 0 | 0
  Participants with Hypertropia: Absence | 25 | 36
  Participants with Hypotropia: Presence | 0 | 0
  Participants with Hypotropia: Absence | 25 | 36

8. Primary Outcome: Number of Participants With Oculomotor Examination (Motility) and Ocular Alignment (Assessed by Corneal Light Reflex and Cover Test) at 24 Months CA
Description: Ocular alignment was assessed in primary gaze by comparing the position of the corneal light reflection in left eye and right eye (corneal light reflection assessment). Presence or absence of strabismus was recorded in primary gaze and in as many of the 9 positions of gaze as feasible with the cover test assessment of refixation movement. Extraocular muscle over action or deficiency was recorded. Ocular motility referred to eye movements governed by the 6 extraocular muscles in each eye. It was assessed by examiner observation of the participants ability to abduct, adduct, supra, and inferoduct each eye. Ocular alignment and motility included the presence or absence of strabismus (classified as Esotropia, Exotropia, Hypertropia, Hypotropia) was recorded. Number of participants with combined data for ocular alignment and oculomotor examination (motility) assessed by corneal light reflex and by the cover test at 24 months CA were reported.
Time Frame: At 24 Months CA
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 34
Participants
  Participants with Esotropia: Presence | 1 | 5
  Participants with Esotropia: Absence | 22 | 29
  Participants with Exotropia: Presence | 0 | 1
  Participants with Exotropia: Absence | 23 | 33
  Participants with Hypertropia: Presence | 0 | 0
  Participants with Hypertropia: Absence | 23 | 34
  Participants with Hypotropia: Presence | 0 | 0
  Participants with Hypotropia: Absence | 23 | 34

9. Primary Outcome: Number of Participants With Oculomotor Examination (Motility) and Ocular Alignment (Assessed by Corneal Light Reflex and Cover Test) at 5-Years CA
Description: Ocular alignment was assessed in primary gaze by comparing the position of the corneal light reflection in left eye and right eye (corneal light reflection assessment). Presence or absence of strabismus was recorded in primary gaze and in as many of the 9 positions of gaze as feasible with the cover test assessment of refixation movement. Extraocular muscle over action or deficiency was recorded. Ocular motility referred to eye movements governed by the 6 extraocular muscles in each eye. It was assessed by examiner observation of the participants ability to abduct, adduct, supra, and inferoduct each eye. Ocular alignment and motility included the presence or absence of strabismus (classified as Esotropia, Exotropia, Hypertropia, Hypotropia) was recorded. Number of participants with combined data for ocular alignment and oculomotor examination (motility) assessed by corneal light reflex and by the cover test at 5-Years CA were reported.
Time Frame: At 5 Years CA
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 14 | 17
Participants
  Participants with Esotropia: Presence | 1 | 1
  Participants with Esotropia: Absence | 13 | 16
  Participants with Exotropia: Presence | 0 | 0
  Participants with Exotropia: Absence | 14 | 17
  Participants with Hypertropia: Presence | 0 | 0
  Participants with Hypertropia: Absence | 14 | 17
  Participants with Hypotropia: Presence | 0 | 0
  Participants with Hypotropia: Absence | 14 | 17

10. Primary Outcome: Number of Participants With Nystagmus at 12 Months CA
Description: Nystagmus was observed during the ocular alignment assessments. Presence and absence of nystagmus was reported at 12 Months CA.
Time Frame: At 12 Months CA
Population: Enrolled set included of all participants for whom written informed consent was obtained for this long-term outcome study. Here, "Overall Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Antecedent rhIGF-1/rhIGFBP-3: Participants who were treated with rhIGF-1/rhIGFBP-3 in study ROPP-2008-01 (NCT01096784) .
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 25 | 36
Participants
  Participants with presence of nystagmus | 1 | 2
  Participants with absence of nystagmus | 24 | 34

11. Primary Outcome: Number of Participants With Nystagmus at 24 Months CA
Description: Nystagmus was observed during the ocular alignment assessments. Presence and absence of nystagmus was reported at 24 Months CA.
Time Frame: At 24 Months CA
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 34
Participants
  Participants with presence of nystagmus | 0 | 2
  Participants with absence of nystagmus | 23 | 32

12. Primary Outcome: Number of Participants With Nystagmus at 5 Years CA
Description: Nystagmus was observed during the ocular alignment assessments. Presence and absence of nystagmus was reported at 5 Years CA.
Time Frame: At 5 Years CA
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 14 | 17
Participants
  Participants with presence of nystagmus | 0 | 2
  Participants with absence of nystagmus | 14 | 15

13. Primary Outcome: Refraction With Cycloplegia as Assessed by Retinoscopy at 6 Months CA
Description: Refraction was a measure of the lens power required for a focused image on the retina. Refraction with cycloplegia was measured and recorded in diopters for each eye individually (left eye and right eye). Refraction with cycloplegia performed as part of the corrective lens determination procedure included measurements of sphere, cylinder, axis, and prism for each individual eye (left eye and right eye). For sphere, the negative values are summarized as 'nearsighted', and the positive values (including sphere of 0.00) are summarized as 'farsighted'.
Time Frame: At 6 Months CA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopter
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 25 | 34
Diopter
  Right Eye: Sphere (Nearsighted): number analyzed (Participants) | 6 | 34
  Right Eye: Sphere (Nearsighted) | -1.833 (1.0916) | -1.417 (1.4216)
  Right Eye: Sphere (Farsighted): number analyzed (Participants) | 21 | 34
  Right Eye: Sphere (Farsighted) | 1.976 (1.2572) | 1.838 (1.3256)
  Right Eye: Cylinder: number analyzed (Participants) | 24 | 33
  Right Eye: Cylinder | 0.875 (0.8534) | 0.932 (0.8801)
  Right Eye: Axis: number analyzed (Participants) | 25 | 33
  Right Eye: Axis | 116.4 (58.03) | 106.0 (52.87)
  Right Eye: Prism: number analyzed (Participants) | 0 | 0
  Left Eye: Sphere (nearsighted): number analyzed (Participants) | 6 | 3
  Left Eye: Sphere (nearsighted) | -1.750 (0.9747) | -1.250 (0.9014)
  Left Eye: Sphere (farsighted): number analyzed (Participants) | 22 | 34
  Left Eye: Sphere (farsighted) | 2.034 (1.2731) | 1.831 (1.3494)
  Left Eye: Cylinder: number analyzed (Participants) | 25 | 33
  Left Eye: Cylinder | 0.820 (0.6395) | 0.962 (0.8341)
  Left Eye: Axis: number analyzed (Participants) | 25 | 33
  Left Eye: Axis | 120.3 (52.27) | 108.8 (54.18)
  Left Eye: Prism: number analyzed (Participants) | 0 | 0

14. Primary Outcome: Refraction With Cycloplegia as Assessed by Retinoscopy at 12 Month CA
Description: as for outcome 13
Time Frame: At 12 Months CA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopter
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 30
Diopter
  Right Eye: Sphere (Nearsighted): number analyzed (Participants) | 7 | 4
  Right Eye: Sphere (Nearsighted) | -1.564 (1.8752) | -2.438 (1.4773)
  Right Eye: Sphere (Farsighted): number analyzed (Participants) | 18 | 27
  Right Eye: Sphere (Farsighted) | 2.042 (1.1796) | 1.491 (1.0908)
  Right Eye: Cylinder: number analyzed (Participants) | 23 | 27
  Right Eye: Cylinder | 0.783 (0.7163) | 0.926 (0.6423)
  Right Eye: Axis | 86.0 (62.82) | 105.7 (50.53)
  Right Eye: Prism: number analyzed (Participants) | 15 | 25
  Right Eye: Prism | 0.00 (0.000) | 0.00 (0.000)
  Left Eye: Sphere (Nearsighted): number analyzed (Participants) | 4 | 5
  Left Eye: Sphere (Nearsighted) | -2.875 (1.9203) | -2.500 (1.7048)
  Left Eye: Sphere (Farsighted): number analyzed (Participants) | 21 | 26
  Left Eye: Sphere (Farsighted) | 1.857 (1.3171) | 1.606 (1.1962)
  Left Eye: Cylinder: number analyzed (Participants) | 23 | 27
  Left Eye: Cylinder | 0.663 (0.6334) | 0.851 (0.6795)
  Left Eye: Axis: number analyzed (Participants) | 22 | 27
  Left Eye: Axis | 107.3 (60.19) | 112.6 (55.11)
  Left Eye: Prism: number analyzed (Participants) | 15 | 25
  Left Eye: Prism | 0.00 (0.000) | 0.00 (0.000)

15. Primary Outcome: Refraction With Cycloplegia as Assessed by Retinoscopy at 20 Month CA
Description: as for outcome 13
Time Frame: At 20 Months CA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopter
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 31
Diopter
  Right Eye: Sphere (Nearsighted): number analyzed (Participants) | 5 | 5
  Right Eye: Sphere (Nearsighted) | -2.350 (2.4083) | -1.700 (1.6808)
  Right Eye: Sphere (Farsighted): number analyzed (Participants) | 18 | 27
  Right Eye: Sphere (Farsighted) | 1.903 (0.9931) | 1.278 (0.8996)
  Right Eye: Cylinder: number analyzed (Participants) | 21 | 27
  Right Eye: Cylinder | 0.750 (0.6755) | 0.778 (0.6841)
  Right Eye: Axis | 105.0 (62.33) | 122.8 (58.69)
  Right Eye: Prism: number analyzed (Participants) | 15 | 22
  Right Eye: Prism | 0.00 (0.000) | 0.00 (0.000)
  Left Eye: Sphere (Nearsighted): number analyzed (Participants) | 3 | 5
  Left Eye: Sphere (Nearsighted) | -3.500 (1.8028) | -2.600 (1.9733)
  Left Eye: Sphere (Farsighted): number analyzed (Participants) | 20 | 27
  Left Eye: Sphere (Farsighted) | 1.800 (1.2237) | 1.389 (1.1080)
  Left Eye: Cylinder: number analyzed (Participants) | 20 | 29
  Left Eye: Cylinder | 0.900 (0.8288) | 0.681 (0.5665)
  Left Eye: Axis: number analyzed (Participants) | 21 | 28
  Left Eye: Axis | 117.8 (53.82) | 110.1 (53.56)
  Left Eye: Prism: number analyzed (Participants) | 16 | 23
  Left Eye: Prism | 0.00 (0.000) | 0.00 (0.000)

16. Primary Outcome: Refraction With Cycloplegia as Assessed by Retinoscopy at 4.75 Years CA
Description: as for outcome 13
Time Frame: At 4.75 Years CA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopter
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 17 | 17
Diopter
  Right Eye: Sphere (Nearsighted): number analyzed (Participants) | 1 | 1
  Right Eye: Sphere (Nearsighted) | -8.500 (NA) — SD is not evaluable for single participants mean data point | -0.500 (NA) — SD is not evaluable for single participants mean data point
  Right Eye: Sphere (Farsighted): number analyzed (Participants) | 17 | 15
  Right Eye: Sphere (Farsighted) | 1.691 (1.1094) | 1.383 (1.5465)
  Right Eye: Cylinder: number analyzed (Participants) | 16 | 17
  Right Eye: Cylinder | 0.593 (0.6505) | 0.603 (0.6254)
  Right Eye: Axis | 99.1 (69.95) | 119.0 (56.05)
  Right Eye: Prism: number analyzed (Participants) | 17 | 14
  Right Eye: Prism | 0.02 (0.075) | 0.00 (0.000)
  Left Eye: Sphere (Nearsighted): number analyzed (Participants) | 1 | 1
  Left Eye: Sphere (Nearsighted) | -6.500 (NA) — SD is not evaluable for single participants mean data point | -0.750 (NA) — SD is not evaluable for single participants mean data point
  Left Eye: Sphere (Farsighted): number analyzed (Participants) | 17 | 15
  Left Eye: Sphere (Farsighted) | 1.853 (1.2376) | 1.517 (1.9966)
  Left Eye: Cylinder: number analyzed (Participants) | 15 | 17
  Left Eye: Cylinder | 0.717 (0.7126) | 0.574 (0.5574)
  Left Eye: Axis: number analyzed (Participants) | 16 | 17
  Left Eye: Axis | 88.6 (65.64) | 114.2 (55.17)
  Left Eye: Prism: number analyzed (Participants) | 15 | 13
  Left Eye: Prism | 0.02 (0.056) | 0.00 (0.000)

17. Primary Outcome: Number of Participants With Stereoacuity as Assessed With the Lang Stereotest At 5 Years CA
Description: Stereoacuity, a measure of depth perception, was assessed using the Lang Stereotest. Number of participants with presence and absence of stereopsis (the ability to perceive depth and 3-dimensional structure) was reported.
Time Frame: At 5 Years CA
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 14 | 17
Participants
  Participants with presence of stereopsis | 13 | 16
  Participants with absence of stereopsis | 1 | 1

18. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Time Frame: From start of study up to end of study (up to 6.5 years)
Population: Safety Set included all participants in the Enrolled Set who have safety follow-up data in this long-term outcome study.
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 36 | 40
Participants | 11 | 9

19. Secondary Outcome: Change From Baseline in Body Weight Z-score
Description: Body weight collected using calibrated scales (type of scale was dependent upon participant's age). Measure recorded to the nearest 0.1 kilogram (kg). Z-score based on participants chronological age and utilizing World Health Organization child growth standards by adjusting age and sex- matched means and standard deviations (norm). Z-score is standard score that gives idea of how far from the mean a data point is. If Z-score is 0, it indicates that the data point's score is identical to the mean score. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Baseline is first assessment in the antecedent study (ROPP-2008-01 [NCT01096784]). Change from baseline in body weight Z-score at 6-month, 12-month, 24-month and 5-year CA were reported.
Time Frame: Baseline, 6 Months CA, 12 Months CA, 24 Months CA and 5 Years CA
Population: Enrolled set included all participants for whom written informed consent was obtained for this long-term outcome study. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 28 | 39
Z-score
  Change at 6 Months CA | 4.40 (1.323) | 4.30 (1.146)
  Change at 12 Months CA: number analyzed (Participants) | 26 | 36
  Change at 12 Months CA | 5.08 (1.300) | 4.88 (1.026)
  Change at 24 Months CA: number analyzed (Participants) | 25 | 36
  Change at 24 Months CA | 5.17 (0.885) | 4.99 (0.983)
  Change at 5 Years CA: number analyzed (Participants) | 19 | 24
  Change at 5 Years CA | 5.80 (1.149) | 5.60 (1.660)

20. Secondary Outcome: Change From Baseline in Height Z-score
Description: Height was measured using Z-score. Z-score was calculated based on the participants chronological age and utilizing World Health Organization child growth standards by adjusting age and sex- matched means and standard deviations (norm). Z-score is a standard score that gives an idea of how far from the mean a data point is. If a Z-score is 0, it indicates that the data point's score is identical to the mean score. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Baseline was defined as the first assessment in the antecedent study (ROPP-2008-01 [NCT01096784]). Change from baseline in Height Z-score at 6-month, 12-month, 24-month and 5-year CA were reported.
Time Frame: Baseline, 6 Months CA, 12 Month CA, 24 Months CA and 5 Years CA
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 28 | 39
Z-Score
  Change at 6 Months CA | 6.36 (1.711) | 6.19 (1.215)
  Change at 12 Months CA: number analyzed (Participants) | 26 | 36
  Change at 12 Months CA | 6.79 (1.747) | 7.25 (1.155)
  Change at 24 Months CA: number analyzed (Participants) | 25 | 36
  Change at 24 Months CA | 7.30 (2.029) | 7.78 (1.376)
  Change at 5 Years CA: number analyzed (Participants) | 19 | 24
  Change at 5 Years CA | 7.84 (1.856) | 8.17 (1.505)

21. Secondary Outcome: Change From Baseline in Head Circumference Z-score
Description: Head circumference measured for all participants using a "lasso" type, non-stretchable measuring tape such as the Lasso-o tape. Z-score calculated based on participants chronological age and utilizing World Health Organization child growth standards by adjusting age, sex matched means and standard deviations (norm).Z-score is standard score that gives idea of how far from mean a data point is. If a Z-score is 0, it indicates that data point's score is identical to mean score. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Baseline was defined as the first assessment in the antecedent study (ROPP-2008-01 [NCT01096784]). Change from baseline in Head Circumference Z-score at 6, 12 and 24-months reported.
Time Frame: Baseline, 6 Months CA, 12 Months CA and 24 Months CA
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 28 | 39
Z-score
  Change at 6 Months CA | 7.61 (1.535) | 7.12 (1.576)
  Change at 12 Months CA: number analyzed (Participants) | 26 | 36
  Change at 12 Months CA | 8.29 (1.472) | 7.83 (1.567)
  Change at 24 Months CA: number analyzed (Participants) | 25 | 35
  Change at 24 Months CA | 8.44 (1.415) | 8.05 (1.692)

22. Secondary Outcome: Change From Baseline (12 Months CA) in Cognitive Development as Assessed by Bayley Scales of Infant and Toddler Development (BSID-III) Composite Scores at 24 Months CA
Description: BSID-III was to assess cognitive, motor, and language skills, and applicable to children aged 1-42 months. There are 5 subscales, cognitive subscale (Ranges: 55-145) stands alone while 2 language subscales (expressive and receptive) combine to make a total language score (Ranges: 47-153) and 2 motor subtests (fine and gross motor) form combined motor scale (Ranges: 46-154). Higher scores represent greater cognitive, language and motor abilities. Positive value indicates improvement and negative value indicate worsening in cognitive development. The 12 Months CA considered as baseline for this outcome measure. Composite scores derived from various sums of subtest scaled scores and scaled to a metric with a mean of 100 and a standard deviation of 15 and range from 40 to 160. Higher values denote stronger skills and abilities in the domain, indicating better outcomes.
Time Frame: Baseline (12 Months CA), 24 Months CA
Population: Enrolled set included all participants for whom written informed consent was obtained for this long-term outcome study. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 32
Score on a scale
  Cognitive Composite Scores: Change at 24 Months CA | 7.0 (18.45) | 6.6 (21.27)
  Language Composite Scores: Change at 24 Months CA | 2.4 (18.73) | -0.9 (15.79)
  Motor Composite Scores: Change at 24 Months CA | 12.2 (23.54) | 10.8 (18.25)

23. Secondary Outcome: Cognitive Development as Assessed by Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV) Full Scale at 5 Years CA
Description: The WPPSI-IV is a measure of general cognitive development in children that has components of both verbal and non-verbal tasks. It is applicable to preschoolers and young children aged 2 years +6 months to 7 years +7 months and is a direct assessment of a child's cognitive skills. The test framework of the WPPSI-IV is organized into five Primary Index sub scales: Verbal Comprehension, Visual Spatial, Fluid Reasoning, Working Memory, and Processing Speed. The Full Scale includes all of the sub scales at the Primary Index scale level, as well as any additional supplemental subtests that may be used to derive the Full Scale IQ. Composite scores are derived from the sum of sub scaled scores with a mean of 100 and a standard deviation of 15. Composite score for Full Scale IQ and subscales (Verbal Comprehension, Visual Spatial, Fluid Reasoning, Working Memory, and Processing Speed) ranges from 40 (extremely low) to 160 (very superior). Data for Full scale IQ was reported here.
Time Frame: At 5 Years CA
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 11 | 14
Scores on a scale | 97.3 (17.28) | 91.6 (14.17)

24. Secondary Outcome: Number of Participants With Abnormal Physical Examination
Description: Physical examination includes general appearance; head and neck, eyes, ears, nose and throat; chest and lungs; endocrine, cardiovascular system, abdomen, genitourinary, skin and musculoskeletal system.
Time Frame: From start of study drug administration up to end of study (up to 6.5 years)
Population: Safety Set included all participants in the Enrolled Set who have safety follow-up data in this long-term outcome study.
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 36 | 40
Participants | 13 | 18

25. Secondary Outcome: Number of Participants Diagnosed With Neurological Examination for Cerebral Palsy (CP) by Neurological Examination at 24 Months CA
Description: A comprehensive neurological examination for the diagnosis of CP was conducted. The Amiel-Tison neurological examination framework was utilized for this assessment and it was conducted by trained medical professionals. Number of Participants diagnosed with CP by neurological examination at 24 Months CA were reported.
Time Frame: At 24 Months CA
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 25 | 37
Participants | 1 | 5

26. Secondary Outcome: Number of Participants With Normal and Abnormal Hearing Screening Status
Description: Number of participants with any hearing status (normal and abnormal) were reported.
Time Frame: At 6 Months CA and 5 Years CA
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 21 | 28
Participants
  At 6 Months CA: Normal Hearing | 20 | 24
  At 6 Months CA: Abnormal Hearing | 1 | 4
  At 5 Years CA: number analyzed (Participants) | 17 | 21
  At 5 Years CA: Normal Hearing | 15 | 20
  At 5 Years CA: Abnormal Hearing | 2 | 1

27. Secondary Outcome: Change From Baseline (6 Months CA) in Child Behavior as Assessed by Vineland Adaptive Behaviour Scales (VABS-II)
Description: The VABS-II was used to measure the personal and social skills of participants serially over time. This test measures the following 4 key domains: Communication, Daily Living Skills, Socialization, and Motor skills. The domains have the same range and directionality as the adaptive behavior composite score (20-160). Higher scores indicate higher level of cognitive ability. A positive change value indicates improvement and negative value indicates worsening in adaptive functioning. The 6 months CA was considered as baseline for this outcome measure. Change from baseline (6 Months CA) in child behavior as assessed by VABS-II adaptive behavior composite was reported here.
Time Frame: Baseline (6 Months CA), 12 Months CA, 24 Months CA, and 5 Year CA
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 22 | 30
Score on a scale
  Change at 12 Months CA: Adaptive Behavior Composite | -0.3 (14.50) | -1.5 (12.41)
  Change at 24 Months CA: Adaptive Behavior Composite: number analyzed (Participants) | 20 | 30
  Change at 24 Months CA: Adaptive Behavior Composite | 7.8 (16.47) | 0.8 (14.89)
  Change at 5 Years CA: Adaptive Behavior Composite: number analyzed (Participants) | 13 | 15
  Change at 5 Years CA: Adaptive Behavior Composite | -3.2 (20.92) | -3.9 (19.86)

28. Secondary Outcome: Number of Participants With Child Behaviour as Assessed by Child Behaviour Checklist (CBCL) Based on T-Score Clinical Categories
Description: The CBCL (1 ½ to 5) was parent-reported outcome measure used to assess behavioral, emotional, and social functioning of toddlers and preschool children aged 18-60 months. It is composed of 99 items rated on Likert scale and includes 7 syndrome scales under 2 domains (Internalizing and Externalizing Problems): Internalizing includes syndromes of Emotionally Reactive, Anxious/Depressed, Somatic Complaints, and Withdrawn. Externalizing includes syndromes of Aggressive Behavior and Attention Problems. The 2 domains of all 7 scales were combined to form total score range of 23 to 100. For each question, raw scores of all subscales are converted to standardized T-scores. Higher T score indicates more behavior problems. For Internalization, Externalization and Total Behavior Problem, T-scores of less than 60 are considered non-clinical, 60-63 are borderline, and 64 or more are considered clinical.
Time Frame: At 24 Months CA and 5 Years CA
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 23 | 34
Participants
  At 24 Months CA: Internalizing: Non-Clinical | 23 | 32
  At 24 Months CA: Internalizing: Borderline | 0 | 0
  At 24 Months CA: Internalizing: Clinical | 0 | 2
  At 5 Years CA: Internalizing: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Internalizing: Non-Clinical | 15 | 15
  At 5 Years CA: Internalizing: Borderline | 1 | 2
  At 5 Years CA: Internalizing: Clinical | 3 | 3
  At 24 Months CA: Externalizing: Non-Clinical | 21 | 32
  At 24 Months CA: Externalizing: Borderline | 1 | 0
  At 24 Months CA: Externalizing: Clinical | 1 | 2
  At 5 Years CA: Externalizing: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Externalizing: Non-Clinical | 16 | 17
  At 5 Years CA: Externalizing: Borderline | 0 | 2
  At 5 Years CA: Externalizing: Clinical | 3 | 1
  At 24 Months CA: Total Behavior Problems: Non-Clinical | 22 | 31
  At 24 Months CA: Total Behavior Problems: Borderline | 1 | 3
  At 24 Months CA: Total Behavior Problems: Clinical | 0 | 0
  At 5 Years CA: Total Behavior Problems: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Total Behavior Problems: Non-Clinical | 14 | 17
  At 5 Years CA: Total Behavior Problems: Borderline | 3 | 2
  At 5 Years CA: Total Behavior Problems: Clinical | 2 | 1

29. Secondary Outcome: Child Behavior as Assessed by Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS) Based on Total Score
Description: The ADHD-RS measures the behaviors of children with Attention-Deficit/Hyperactivity Disorder (ADHD). It consisted of 18 items designed to reflect current symptomatology of ADHD based on DSM-IV criteria. Each item was scored on a 4-point scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0 to 54. Higher scores represent greater severity of ADHD symptoms.
Time Frame: At 5 Years CA
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 18 | 20
Score on scale | 11.9 (9.30) | 8.3 (10.10)

30. Secondary Outcome: Child Behavior as Assessed by Social Communication Questionnaire (SCQ)
Description: The SCQ is a brief instrument evaluate communication skills and social functioning in children used for screening for autism or autism spectrum disorders (ASD). The SCQ has 40 dichotomous (yes, no) items, and each item scored 1 point for "abnormal behavior" and 0 point for "absence of abnormal behavior/normal behavior." It yields total score ranging from 0 to 39, higher scores represent more social communication impairment. The first item, "Is she/he now able to talk using short phrases or sentences?", is not scored, but determines if six items relating to abnormal language are assigned. Only "verbal" children (children with "yes" response to first question) are assigned the six items relating to abnormal language and can score a total of 0 to 39 points; "non-verbal" children (children with "no" response to first question) are not assigned six items in relation to abnormal language and score a total of 0 to 33 points where higher scores represent more social communication impairment.
Time Frame: At 5 Years CA
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 19 | 20
Score on scale | 5.9 (6.80) | 5.2 (7.88)

31. Secondary Outcome: Number of Participants With Pulmonary Morbidity
Description: Pulmonary morbidity was assessed with questions related to family history and smoking status as well as diagnosis of select pulmonary symptoms, conditions and related hospitalizations. Anyone living in the same home with participant smoke, Participants had asthma, wheezing, bronchopulmonary dysplasia (BPD) exacerbation or flare-up, Participants had bronchiolitis, bronchitis, or pneumonia diagnosed, Participants had to use oxygen at home, Participants had to visit emergency room or urgent care for respiratory problem, and Participants had to stay in a hospital overnight for respiratory problem were reported.
Time Frame: At 6 Months CA, 12 Months CA and 24 Months CA
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 28 | 39
Participants
  At 6 Months CA: Anyone living in the same home with participant smoke: Yes | 6 | 7
  At 6 Months CA: Anyone living in the same home with participant smoke: No | 22 | 32
  At 6 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: Yes | 8 | 4
  At 6 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: No | 20 | 35
  At 6 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: Yes | 4 | 5
  At 6 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: No | 24 | 34
  At 6 Months CA: Had to use oxygen at home: Yes | 8 | 5
  At 6 Months CA: Had to use oxygen at home: No | 20 | 34
  At 6 Months CA: Had to visit emergency room or urgent care for respiratory problem: Yes | 5 | 7
  At 6 Months CA: Had to visit emergency room or urgent care for respiratory problem: No | 23 | 32
  At 6 Months CA: Had to stay in a hospital overnight for respiratory problem: Yes | 5 | 7
  At 6 Months CA: Had to stay in a hospital overnight for respiratory problem: No | 23 | 32
  At 12 Months CA: Anyone living in the same home with participant smoke: number analyzed (Participants) | 26 | 35
  At 12 Months CA: Anyone living in the same home with participant smoke: Yes | 3 | 5
  At 12 Months CA: Anyone living in the same home with participant smoke: No | 23 | 30
  At 12 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: number analyzed (Participants) | 26 | 35
  At 12 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: Yes | 4 | 7
  At 12 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: No | 22 | 28
  At 12 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: number analyzed (Participants) | 26 | 35
  At 12 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: Yes | 1 | 5
  At 12 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: No | 25 | 30
  At 12 Months CA: Had to use oxygen at home: number analyzed (Participants) | 26 | 35
  At 12 Months CA: Had to use oxygen at home: Yes | 2 | 0
  At 12 Months CA: Had to use oxygen at home: No | 24 | 35
  At 12 Months CA: Had to visit emergency room or urgent care for respiratory problem: number analyzed (Participants) | 26 | 35
  At 12 Months CA: Had to visit emergency room or urgent care for respiratory problem: Yes | 3 | 7
  At 12 Months CA: Had to visit emergency room or urgent care for respiratory problem: No | 23 | 28
  At 12 Months CA: Had to stay in a hospital overnight for respiratory problem: number analyzed (Participants) | 26 | 35
  At 12 Months CA: Had to stay in a hospital overnight for respiratory problem: Yes | 1 | 4
  At 12 Months CA: Had to stay in a hospital overnight for respiratory problem: No | 25 | 31
  At 24 Months CA: Anyone living in the same home with participant smoke: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Anyone living in the same home with participant smoke: Yes | 3 | 3
  At 24 Months CA: Anyone living in the same home with participant smoke: No | 22 | 33
  At 24 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: Yes | 4 | 8
  At 24 Months CA: Had asthma, wheezing, BPD exacerbation or flare-up: No | 21 | 28
  At 24 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: Yes | 2 | 1
  At 24 Months CA: Had bronchiolitis, bronchitis, or pneumonia diagnosed: No | 23 | 35
  At 24 Months CA: Had to use oxygen at home: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Had to use oxygen at home: Yes | 1 | 0
  At 24 Months CA: Had to use oxygen at home: No | 24 | 36
  At 24 Months CA: Had to visit emergency room or urgent care for respiratory problem: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Had to visit emergency room or urgent care for respiratory problem: Yes | 5 | 5
  At 24 Months CA: Had to visit emergency room or urgent care for respiratory problem: No | 20 | 31
  At 24 Months CA: Had to stay in a hospital overnight for respiratory problem: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Had to stay in a hospital overnight for respiratory problem: Yes | 2 | 0
  At 24 Months CA: Had to stay in a hospital overnight for respiratory problem: No | 23 | 36

32. Secondary Outcome: Number of Participants With Survival Status
Description: Survival status was assessed by number participants who died and were censored during the study.
Time Frame: From start of study drug administration up to end of study (up to 6.5 years)
Population: Safety set included all participants in the Enrolled Set who have safety follow-up data in this long-term outcome study.
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 36 | 40
Participants
  Participants who Died | 1 | 0
  Participants who were Censored | 35 | 40

33. Secondary Outcome: Change From Baseline (3 Months CA) in Pediatric Quality of Life Inventory (PedsQL™) Scale: Infant Scale
Description: The PedsQL was a generic health related quality of life instrument designed specifically for a pediatric population. PedsQL infant scale encompasses 5 dimensions of functioning (Physical Functioning, Physical Symptoms, Emotional Functioning, Social Functioning, and Cognitive Functioning). The infant for ages 1-12 months (36 Items); for ages 13-24 months (45 Items) rated on a 5-point Likert scale (0 to 4). Overall total scores were calculated as average of all dimensional sub-score items of Infant scale, ranging from 0 to 100 where 0=100 (Never), 1=75 (almost never), 2=50 (sometimes), 3=25 (often), and 4=0 (almost always). Higher scores indicate improved quality of life. A negative value indicates decreased quality of life. The 3 months CA was considered as baseline for this outcome measure.
Time Frame: Baseline (3 Months CA) up to 6 Months CA, 12 Months CA and 24 Months CA
Population: Enrolled set included all participants for whom written informed consent was obtained for this long-term outcome study. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 28 | 38
Score on scale
  Change at 6 Months CA: Total Score (Infant scale) | -1.10 (10.056) | -0.60 (11.088)
  Change at 12 Months CA: Total Score (Infant scale): number analyzed (Participants) | 25 | 36
  Change at 12 Months CA: Total Score (Infant scale) | -0.16 (12.875) | -0.57 (11.902)
  Change at 24 Months CA: Total Score (Infant scale): number analyzed (Participants) | 3 | 7
  Change at 24 Months CA: Total Score (Infant scale) | 7.84 (7.339) | -4.82 (14.205)

34. Secondary Outcome: Change From Baseline (24 Months CA) in Pediatric Quality of Life Inventory (PedsQL™) Scale: Generic Core Scale (GCS) Total Score
Description: The PedsQL was a generic health related quality of life instrument designed specifically for a pediatric population. The GCS encompasses 4 dimensions of functioning (physical, emotional, social, school). The GCS that apply to toddler for 2-4 years of age (21 Items) rated on a 5-point Likert scale (0 to 4); and Young Child for 5-7 years of age (23 Items) rated on a 3-point Likert scale (0, 2, 4). Overall total scores were calculated as average of all dimensional sub-score items of GCS (Toddler and young children's) ranging from 0 to 100 where 0=100 (Never), 1=75 (almost never), 2=50 (sometimes), 3=25 (often), and 4=0 (almost always). Higher scores indicate improved quality of life. A negative value indicates decreased quality of life. The 24 month CA was considered as baseline for this outcome measure.
Time Frame: Baseline (24 Months CA), up to 3 Years CA, 4 Years CA and 5 Years CA
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 19 | 22
Score on scale
  Change at 3 Years CA: Total Score | 0.62 (12.220) | -1.13 (8.533)
  Change at 4 Years CA: Total Score: number analyzed (Participants) | 19 | 18
  Change at 4 Years CA: Total Score | 1.50 (14.376) | -3.46 (7.917)
  Change at 5 Years CA: Total Score: number analyzed (Participants) | 16 | 15
  Change at 5 Years CA: Total Score | -4.96 (15.561) | -4.49 (8.225)

35. Secondary Outcome: Number of Participants With Health Status Measured by the Health Status Classification System-Preschool (HSCS-PS)
Description: HSCS-PS was a validated instrument used via parent proxy within age 2.5 - 5 years. The instrument is composed of 12 domains (Vision, Hearing, Speech, Mobility, Dexterity, Self-care, Emotion, Learn/Remember, Think/Problem Solve, Pain, General Health, Behavior) with up to 6 levels (0-5). The 12 dimensions grouped into 4 categories: neurosensory (vision and hearing), motor (mobility, dexterity, and self-care), learning/remembering (speech, learn/remember, think/problem solve), and quality of life (emotion, pain, general health, behavior). For each category, data were recorded into following levels: no problem (scoring 0 on any attribute); a mild problem (scoring 1 on a scale of 0 to 3, or 1 to 2 on a scale of 0 to 5 for any attribute);moderate/severe problem (scoring > 1 on a scale of 0 to 3, or >2 on a scale of 0 to 5 for any attribute). Higher numbers indicating better child's health status.
Time Frame: At 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 24 | 35
Participants
  At 24 Months CA: Neurosensory: No Problem | 21 | 30
  At 24 Months CA: Neurosensory: Mild | 3 | 4
  At 24 Months CA: Neurosensory: Moderate/Severe | 0 | 1
  At 24 Months CA: Motor: No Problem | 19 | 21
  At 24 Months CA: Motor: Mild | 3 | 9
  At 24 Months CA: Motor: Moderate/Severe | 2 | 5
  At 24 Months CA: Learning/Remembering: No Problem | 10 | 10
  At 24 Months CA: Learning/Remembering: Mild | 6 | 13
  At 24 Months CA: Learning/Remembering: Moderate/Severe | 8 | 12
  At 24 Months CA: Quality of Life: No Problem | 11 | 21
  At 24 Months CA: Quality of Life: Mild | 11 | 11
  At 24 Months CA: Quality of Life: Moderate/Severe | 2 | 3
  At 3 Years CA: Neurosensory: number analyzed (Participants) | 24 | 33
  At 3 Years CA: Neurosensory: No Problem | 20 | 28
  At 3 Years CA: Neurosensory: Mild | 2 | 3
  At 3 Years CA: Neurosensory: Moderate/Severe | 2 | 2
  At 3 Years CA: Motor: number analyzed (Participants) | 24 | 33
  At 3 Years CA: Motor: No Problem | 16 | 16
  At 3 Years CA: Motor: Mild | 4 | 13
  At 3 Years CA: Motor: Moderate/Severe | 4 | 4
  At 3 Years CA: Learning/Remembering: number analyzed (Participants) | 24 | 33
  At 3 Years CA: Learning/Remembering: No Problem | 13 | 17
  At 3 Years CA: Learning/Remembering: Mild | 6 | 11
  At 3 Years CA: Learning/Remembering: Moderate/Severe | 5 | 5
  At 3 Years CA: Quality of Life: number analyzed (Participants) | 24 | 33
  At 3 Years CA: Quality of Life: No Problem | 13 | 21
  At 3 Years CA: Quality of Life: Mild | 9 | 8
  At 3 Years CA: Quality of Life: Moderate/Severe | 2 | 4
  At 4 Years CA: Neurosensory: number analyzed (Participants) | 23 | 27
  At 4 Years CA: Neurosensory: No Problem | 21 | 23
  At 4 Years CA: Neurosensory: Mild | 2 | 4
  At 4 Years CA: Neurosensory: Moderate/Severe | 0 | 0
  At 4 Years CA: Motor: number analyzed (Participants) | 23 | 27
  At 4 Years CA: Motor: No Problem | 16 | 16
  At 4 Years CA: Motor: Mild | 5 | 8
  At 4 Years CA: Motor: Moderate/Severe | 2 | 3
  At 4 Years CA: Learning/Remembering: number analyzed (Participants) | 23 | 27
  At 4 Years CA: Learning/Remembering: No Problem | 16 | 12
  At 4 Years CA: Learning/Remembering: Mild | 4 | 11
  At 4 Years CA: Learning/Remembering: Moderate/Severe | 3 | 4
  At 4 Years CA: Quality of Life: number analyzed (Participants) | 23 | 27
  At 4 Years CA: Quality of Life: No Problem | 13 | 17
  At 4 Years CA: Quality of Life: Mild | 8 | 9
  At 4 Years CA: Quality of Life: Moderate/Severe | 2 | 1
  At 5 Years CA: Neurosensory: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Neurosensory: No Problem | 16 | 17
  At 5 Years CA: Neurosensory: Mild | 3 | 3
  At 5 Years CA: Neurosensory: Moderate/Severe | 0 | 0
  At 5 Years CA: Motor: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Motor: No Problem | 13 | 14
  At 5 Years CA: Motor: Mild | 5 | 5
  At 5 Years CA: Motor: Moderate/Severe | 1 | 1
  At 5 Years CA: Learning/Remembering: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Learning/Remembering: No Problem | 10 | 12
  At 5 Years CA: Learning/Remembering: Mild | 7 | 7
  At 5 Years CA: Learning/Remembering: Moderate/Severe | 2 | 1
  At 5 Years CA: Quality of Life: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Quality of Life: No Problem | 11 | 15
  At 5 Years CA: Quality of Life: Mild | 8 | 4
  At 5 Years CA: Quality of Life: Moderate/Severe | 0 | 1

36. Secondary Outcome: Health Status Measured by the Health Utilities Index (HUI) Mark 2 and 3
Description: The HUI is a family of generic health profiles and preference-based systems used for measuring health status, reporting HRQoL, and producing utility scores. The HUI2 score includes 6 attributes: Sensation, Mobility, Cognition, Self-Care, Emotion, and Pain with up to 5 levels of severity (higher numbers indicate worse level of severity). The HUI3 score includes 8 attributes: Vision, Hearing, Speech, Cognition, Ambulation, Dexterity, Emotion, and Pain with up to 6 levels to indicate the severity (with higher numbers indicating worse levels). HUI2/3 single-attribute scores of morbidities are defined on a scale such the worst level has a score of 0.00 and the best level has a score of 1.00. HUI mark 2 and 3 Overall utility score was reported.
Time Frame: At 5 Years CA
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 19 | 20
Score on scale
  HUI2 Overall Utility Score | 0.929 (0.1246) | 0.867 (0.2115)
  HUI3 Overall Utility Score | 0.893 (0.1960) | 0.852 (0.2665)

37. Secondary Outcome: Health Care Resource Use (HCRU)
Description: The total number of private office/hospital outpatient visits of health care resource at 3 Months CA, 6 Months CA, 12 Months CA, 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA were reported.
Time Frame: At 3 Months CA, 6 Months CA, 12 Months CA, 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 29 | 39
Visits
  At 3 Months CA: Total Health Care Resource Use | 9.8 (6.48) | 8.3 (7.67)
  At 6 Months CA: Total Health Care Resource Use: number analyzed (Participants) | 28 | 37
  At 6 Months CA: Total Health Care Resource Use | 15.5 (16.06) | 10.3 (9.40)
  At 12 Months CA: Total Health Care Resource Use: number analyzed (Participants) | 25 | 36
  At 12 Months CA: Total Health Care Resource Use | 25.0 (23.81) | 22.5 (33.95)
  At 24 Months CA: Total Health Care Resource Use: number analyzed (Participants) | 25 | 35
  At 24 Months CA: Total Health Care Resource Use | 20.1 (31.95) | 30.0 (40.92)
  At 3 Years CA: Total Health Care Resource Use: number analyzed (Participants) | 24 | 31
  At 3 Years CA: Total Health Care Resource Use | 22.8 (41.38) | 34.8 (55.25)
  At 4 Years CA: Total Health Care Resource Use: number analyzed (Participants) | 20 | 23
  At 4 Years CA: Total Health Care Resource Use | 21.8 (39.00) | 41.2 (69.93)
  At 5 Years CA: Total Health Care Resource Use: number analyzed (Participants) | 16 | 15
  At 5 Years CA: Total Health Care Resource Use | 15.7 (39.80) | 32.7 (51.22)

38. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits to Emergency Department
Description: Number of visits to emergency department at 3 Months CA, 6 Months CA, 12 Months CA, 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA were reported.
Time Frame: At 3 Months CA, 6 Months CA, 12 Months CA , 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 15 | 17
Visits
  At 3 Months CA: Emergency Department Visits: number analyzed (Participants) | 6 | 7
  At 3 Months CA: Emergency Department Visits | 2.5 (1.87) | 1.6 (1.13)
  At 6 Months CA: Emergency Department Visits: number analyzed (Participants) | 5 | 10
  At 6 Months CA: Emergency Department Visits | 2.2 (2.17) | 1.3 (0.67)
  At 12 Months CA: Emergency Department Visits: number analyzed (Participants) | 9 | 13
  At 12 Months CA: Emergency Department Visits | 1.6 (0.73) | 2.2 (1.14)
  At 24 Months CA: Emergency Department Visits | 2.1 (1.39) | 1.4 (0.61)
  At 3 Years CA: Emergency Department Visits: number analyzed (Participants) | 11 | 14
  At 3 Years CA: Emergency Department Visits | 2.5 (2.38) | 1.6 (0.84)
  At 4 Years CA: Emergency Department Visits: number analyzed (Participants) | 7 | 6
  At 4 Years CA: Emergency Department Visits | 1.9 (1.46) | 1.7 (0.82)
  At 5 Years CA: Emergency Department Visits: number analyzed (Participants) | 3 | 1
  At 5 Years CA: Emergency Department Visits | 1.7 (0.58) | 1 (NA) — SD is not evaluable for single mean data point.

39. Secondary Outcome: Health Care Resource Utilization (HCRU): Duration of Hospitalization
Description: The participant's duration of hospitalizations at 3 Months CA, 6 Months CA, 12 Months CA, 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA were reported.
Time Frame: At 3 Months CA, 6 Months CA, 12 Months CA , 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 9 | 12
Days
  At 3 Months CA: number analyzed (Participants) | 9 | 11
  At 3 Months CA | 12.9 (31.27) | 5.5 (4.55)
  At 6 Months CA | 6.4 (4.56) | 7.4 (9.58)
  At 12 Months CA: number analyzed (Participants) | 5 | 9
  At 12 Months CA | 7.2 (7.76) | 9.0 (11.87)
  At 24 Months CA: number analyzed (Participants) | 7 | 4
  At 24 Months CA | 4.1 (5.01) | 2.5 (1.73)
  At 3 Years CA: number analyzed (Participants) | 4 | 5
  At 3 Years CA | 4.3 (3.30) | 4.8 (6.87)
  At 4 Years CA: number analyzed (Participants) | 2 | 3
  At 4 Years CA | 3.5 (3.54) | 4.0 (3.61)
  At 5 Years CA: number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Required Prescription Eyeglasses and Educational Support
Description: Number of participants who required prescription eyeglasses and educational support at 3 Months CA, 6 Months CA, 12 Months CA, 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA were reported.
Time Frame: At 3 Months CA, 6 Months CA, 12 Months CA, 24 Months CA, 3 Years CA, 4 Years CA and 5 Years CA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
Number analyzed (Participants) | 32 | 39
Participants
  At 3 Months CA: Used Prescription Eyeglasses: Yes | 0 | 0
  At 3 Months CA: Used Prescription Eyeglasses: No | 32 | 39
  At 6 Months CA: Used Prescription Eyeglasses: number analyzed (Participants) | 28 | 39
  At 6 Months CA: Used Prescription Eyeglasses: Yes | 0 | 0
  At 6 Months CA: Used Prescription Eyeglasses: No | 28 | 39
  At 12 Months CA: Used Prescription Eyeglasses: number analyzed (Participants) | 26 | 36
  At 12 Months CA: Used Prescription Eyeglasses: Yes | 0 | 1
  At 12 Months CA: Used Prescription Eyeglasses: No | 26 | 35
  At 24 Months CA: Used Prescription Eyeglasses: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Used Prescription Eyeglasses: Yes | 1 | 2
  At 24 Months CA: Used Prescription Eyeglasses: No | 24 | 34
  At 3 Years CA: Used Prescription Eyeglasses: number analyzed (Participants) | 24 | 33
  At 3 Years CA: Used Prescription Eyeglasses: Yes | 3 | 7
  At 3 Years CA: Used Prescription Eyeglasses: No | 21 | 26
  At 4 Years CA: Used Prescription Eyeglasses: number analyzed (Participants) | 23 | 27
  At 4 Years CA: Used Prescription Eyeglasses: Yes | 2 | 5
  At 4 Years CA: Used Prescription Eyeglasses: No | 21 | 22
  At 5 Years CA: Used Prescription Eyeglasses: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Used Prescription Eyeglasses: Yes | 3 | 4
  At 5 Years CA: Used Prescription Eyeglasses: No | 16 | 16
  At 3 Months CA: Received Educational Support: Yes | 0 | 0
  At 3 Months CA: Received Educational Support: No | 32 | 39
  At 6 Months CA: Received Educational Support: number analyzed (Participants) | 28 | 39
  At 6 Months CA: Received Educational Support: Yes | 0 | 1
  At 6 Months CA: Received Educational Support: No | 28 | 38
  At 12 Months CA: Received Educational Support: number analyzed (Participants) | 26 | 36
  At 12 Months CA: Received Educational Support: Yes | 0 | 1
  At 12 Months CA: Received Educational Support: No | 26 | 35
  At 24 Months CA: Received Educational Support: number analyzed (Participants) | 25 | 36
  At 24 Months CA: Received Educational Support: Yes | 0 | 0
  At 24 Months CA: Received Educational Support: No | 25 | 36
  At 3 Years CA: Received Educational Support: number analyzed (Participants) | 24 | 33
  At 3 Years CA: Received Educational Support: Yes | 1 | 4
  At 3 Years CA: Received Educational Support: No | 23 | 29
  At 4 Years CA: Received Educational Support: number analyzed (Participants) | 23 | 27
  At 4 Years CA: Received Educational Support: Yes | 5 | 3
  At 4 Years CA: Received Educational Support: No | 18 | 24
  At 5 Years CA: Received Educational Support: number analyzed (Participants) | 19 | 20
  At 5 Years CA: Received Educational Support: Yes | 3 | 5
  At 5 Years CA: Received Educational Support: No | 16 | 15

ADVERSE EVENTS:
Time Frame: From start of study up to end of the study (up to 6.5 years)
Arm/Group | Antecedent Standard of Care | Antecedent rhIGF-1/rhIGFBP-3
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/40
Serious Adverse Events (participants affected / at risk) | 3/36 | 2/40
Other Adverse Events (participants affected / at risk) | 5/36 | 2/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antecedent Standard of Care (N=36) | Antecedent rhIGF-1/rhIGFBP-3 (N=40)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antecedent Standard of Care (N=36) | Antecedent rhIGF-1/rhIGFBP-3 (N=40)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT02386839/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT02386839/SAP_001.pdf